CLINICAL TRIAL: NCT05123378
Title: Assessing the Impact of the Liberia National Community Health Assistant (NCHA) Program on Under-five Mortality: A Study Protocol
Brief Title: Liberia National Community Health Assistant (NCHA) Program and Under-five Mortality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Last Mile Health (Other)
Collaborators: Heidelberg University (Other); Northwestern University (Other); Georgetown University (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro00048901
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Malaria; Diarrhea; Acute Respiratory Infection; Malnutrition, Child
Keywords: Community Health; Mortality; Health Care Utilization; Child Illness Prevalence; Experiential Quality
MeSH Terms: conditions — Malaria; Diarrhea; Child Nutrition Disorders; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: The NCHAP is being implemented in Grand Bassa county on a staggered schedule across eight study districts between 2018 and 2022. In order to serve most indigent districts first, the order is not randomized. Districts with more need for health interventions have been prioritized in the implementation roll out. All program implementations are preceded by community engagement activities, especially in getting the involvement of political and traditional leaders in the community and a training period for CHWs of a few months. Within this time CHWs are recruited and trained in a modular approach with in class training followed by practice in the community for mastery before the next module. The implementation process is still ongoing and the NCHA program will continue after the end of the study in 2022.
Masking Description: All participants, care providers, investigators, and outcome assessors are aware of where and when the intervention is being delivered in each community in Grand Bassa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1 Implementation (Experimental): Campwood District and District 3C begin NCHAP implementation in May 2018.
  Interventions: Behavioral: Liberia National Community Health Assistant Program
- Phase 2 Implementation (Experimental): District 3AB and District 2 begin NCHAP implementation in November 2018.
  Interventions: Behavioral: Liberia National Community Health Assistant Program
- Phase 3 Implementation (Experimental): District 4 begins NCHAP implementation in September 2020.
  Interventions: Behavioral: Liberia National Community Health Assistant Program
- Phase 4 Implementation (Experimental): Owensgrove District and Commonwealth District begin NCHAP implementation in April 2021.
  Interventions: Behavioral: Liberia National Community Health Assistant Program
- Phase 5 Implementation (Experimental): District 1 begins NCHAP implementation in January 2022.
  Interventions: Behavioral: Liberia National Community Health Assistant Program

INTERVENTIONS:
Behavioral: Liberia National Community Health Assistant Program — Through the National Community Health Assistant Program (NCHAP), members of remote communities select Community Health Assistants (CHAs). Once selected, CHAs are trained to deliver direct services which include; treatment of diarrhea, ARI, and malaria following Integrated Community Case Management (iCCM) protocols, referrals for patients with clinical danger signs, family planning for women of childbearing age and birth preparedness and education for pregnant women. CHAs are also trained to deliver indirect services which include; health education, active surveillance, referral for mental health and other special conditions for all age groups. Since 2020 COVID-education has also been included in the CHAs work.

SUMMARY:
Last Mile Health (LMH) has partnered with the Liberian Ministry of Health (MOH) to support the design and implementation of the National Community Health Assistant Program (NCHAP). In collaboration with MOH, LMH is planning to conduct an impact evaluation in Grand Bassa to assess the effect of the National Community Health Assistant Program (NCHAP) on health outcomes, as well as to learn lessons around program operations and implementation. Our central hypothesis is that Community Health Assistants (CHAs) within the NCHAP will reduce under 5 mortality, as a result of expanding access to and uptake of health care utilization in remote communities. We will use a mixed effects discrete survival model, taking advantage of the staggered program implementation in Grand Bassa districts over a period of 4 years to compare the incidence of under-5 child mortality between the pre- and post-CHW program implementation periods.

DETAILED DESCRIPTION:
Previous evaluations of the NCHAP in Rivercess and Grand Gedeh counties found significant increases in uptake of child and maternal health-care services from qualified providers. We will expand upon those studies to assess the impact of the CHA program after a phased implementation in an additional county.

The Liberian NCHAP is being rolled out staggered across the eight districts of Grand Bassa County by the government of Liberia. The practical program implementation is accompanied and supported by LMH. Starting with program implementation in March 2018, the last district will be covered by the NCHAP by January 2022. At baseline, midline, and endline LMH will conduct representative household surveys to assess the interventions uptake and effectiveness on population health. This programmatic strategy allows us to apply a effectiveness-implementation hybrid design, where we are using quasi experimental methods on the intervention's impact on relevant outcomes and program utilization and mixed methods to assess the implementation process.

The program implementation and data collection takes place in the Grand Bassa county of Liberia between 2018 and 2022. Measuring an area of 7,936 square kilometres and an overall population of 224,839 in 2008, the county is predominantly rural. For program roll out the five administrative districts were subdivided in eight study districts (see Figure 1). The target population of the NCHA are households in communities with a distance of more than 5 km from the nearest health facility. According to the 2018 LMH Grand Bassa household survey, 1,733 communities were identified as remote with 23,702 households.

The long-term objective of the NCHA program is to provide community-based health care that substantially improves population health and is desirable and respectful to the clients it serves. In pursuit of this objective, our specific research aims for the Grand Bassa causal impact evaluation is to assess the impact of the NCHA program on under-5 mortality.

ELIGIBILITY:
The intervention will be accessable for everyone in the target communities without eligbilty criteria.

The impact assessment survey will be a full census. All remote target communities in Grand Bassa will be selected and all households within selected communities will be surveyed with the child mortality module and for other core indicators. Within each household the survey population will consist of all women of reproductive age who are at least 15 years old (15-49). We will select all 1,733 remote communities in the study area of Grand Bassa covering 23,702 households.

Inclusion Criteria:

* Communities >5 km from a health facility
* Within a household all women 18-49 were interviewed (if possible).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23702 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Mortality in children under 5 | Cross-sectional household surveys administered at endline in 2022
  Assess the impact of the NCHA program on under-5 mortality

SECONDARY OUTCOMES:
Health care utilization | Cross-sectional household surveys administered at baseline in 2018, midline 2019 and 2021, and endline in 2022
  Determine effects of the NCHA program on health care utilization
Child illness prevalence | Cross-sectional household surveys administered at baseline in 2018, midline 2019 and 2021, and endline in 2022
  Determine effects of the NCHA program on child illness prevalence
Experiential quality and trust in the health care system | Cross-sectional household surveys administered at baseline in 2018, midline 2019 and 2021, and endline in 2022
  Determine effects of the NCHA program on experiential quality and trust in the health care system

CONTACTS AND LOCATIONS:
Overall Officials: Marion Subah, Principal Investigator — marionsubah@lastmilehealth.org
Locations (1):
- Last Mile Health, Monrovia, Montserrado County, Liberia

IPD SHARING:
Plan to Share IPD: No
Requests can be made of the PI.